CLINICAL TRIAL: NCT03879018
Title: Retraining Reaching in Cerebellar Ataxia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amy J. Bastian, Ph.D., Professor of Neuroscience, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00182673; 2R01HD040289-15A1 (NIH)
Record Dates: First submitted 2019-03-08; First posted 2019-03-18 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cerebellar Ataxia
Keywords: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Feedback, Sensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reinforcement Training (Experimental): Reach training with visual feedback. During each training session, participants will first be familiarized with the task and then will reach from a home position to 4 virtual targets that are presented in the front of the participant and within the workspace where most natural arm movements are performed. During training the participant will reach a total of 400 times. For reinforcement training, participants will not see their hand or a cursor, but instead participants will receive target-specific binary feedback after each reach (i.e. based on running average of last 10 reaches to that target). Binary feedback indicates only whether the reach was successful or unsuccessful and provides no specific information about the location of the hand.
  Interventions: Behavioral: Reach training with visual feedback
- Standard Practice Training (Experimental): Reach training with visual feedback. During each training session, participants will first be familiarized with the task and then will reach from a home position to 4 virtual targets that are presented in the front of the participant and within the workspace where most natural arm movements are performed. During training the participant will reach a total of 400 times. For standard practice, participants will be able to see a cursor that represents the position of the hand at all times and try to make straight reaches to the targets. This type of feedback provided specific information about the location of the hand.
  Interventions: Behavioral: Reach training with visual feedback

INTERVENTIONS:
Behavioral: Reach training with visual feedback — Reach training will be accomplished using an Oculus Rift and Touch 3D headset. Active markers will be placed on the shoulder, elbow, wrist, and finger in order to capture limb movement in real time. During each training session, participants will first be familiarized with the task and then will reach from a home position to 4 virtual targets that are presented in the front of the participant and within the workspace where most natural arm movements are performed.Targets will be presented in a pseudorandom order and participants will reach a total of 400 times

SUMMARY:
The purpose of this study is to test for benefits of reinforcement based training paradigm versus standard practice over weeks for improving reaching movements in people with ataxia.

DETAILED DESCRIPTION:
Damage to the cerebellum produces characteristic deficits in movement coordination, known as "ataxia." Reaching movements become curved, tremulous, and over- or undershoot targets, thus affecting nearly all activities of daily living. Sitting and standing balance becomes unsteady, and walking has a characteristic 'drunken' appearance with lateral veering and a widening of the base of support. People with many types of neurological diseases (e.g. autosomal dominant ataxias (e.g. SCAs), multiple sclerosis, cerebral palsy, stroke, Freidreich's ataxia) often have disabling ataxia.

In past work the investigators have shown that many individuals with ataxia from cerebellar disease can learn simple visuomotor tasks using reinforcement learning paradigms. The investigators do not know if individuals with ataxia from cerebellar disease can improve more complex motor patterns. In general, there are few rehabilitation studies on ataxia, with most focusing on balance and walking. Yet, arm ataxia is a significant problem that affects most all activities of daily living (e.g. eating, cooking, bathing, dressing, working). Many studies have assessed reaching ataxia on single days in order to try to better understand the fundamental basis for ataxic arm movements. Based on previous literary searches, there are only a couple of small studies that have tested whether training over weeks can mitigate arm ataxia. Each of these was a case series of either 3 or 4 people, and all patients had ataxia from lesions that included structures outside of the cerebellum. Both showed some positive effects but responses varied across patients. This work that the investigators propose will look at the affects of a longer training regimen of upper limb reaching in people with cerebellar ataxia.

The investigators will study cerebellar patients that have shown the ability to learn from previous work. Subjects with cerebellar ataxia will be randomized into two groups to receive either reinforcement training or standard practice training over a 12 week period. Subjects will train for 45 minutes a day, 3 times per week for two weeks for each type of training, with a two week 'rest' period in between. After training, subjects will be asked to return for two visits to test for retention. On each training day, reinforcement training (or standard practice) will be done using an Oculus Rift and Touch 3D headset. Training encompasses reaching to a 3D target with either online visual feedback or binary feedback 400 times. Motion tracking sensors will be placed on the shoulder, elbow, wrist, and finger, in order to track movement data in real time. These studies will provide important new information about upper limb long term training with visual feedback in individuals with Cerebellar Ataxia

ELIGIBILITY:
Inclusion Criteria:

* Cerebellar damage from stroke, tumor or degeneration
* Age 22-80

Exclusion Criteria:

* Clinical or MRI evidence of damage to extracerebellar brain (e.g. multiple system atrophy)
* Extrapyramidal symptoms, peripheral vestibular loss, or sensory neuropathy
* Dementia ( Mini-Mental State exam > 22)
* Pain that interferes with the tasks
* Vision loss that interferes with the tasks

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Hand path distance during natural reaching to the trained target locations. | Assessed every study visit week 1 to week 12
  Hand path distance is the percent above an ideal (straight reach) averaged over reaches to all 4 targets. To collect this measure, investigators will use motion capture equipment to record the positions of active markers that subjects will wear on their shoulder, elbow, wrist, and finger.

SECONDARY OUTCOMES:
ICARS (International Cooperative Ataxia Rating Scale) | Assessed week 1 before the first training session, and week 12
  ICARS is a standardized scale used to quantify the level of impairment in people with cerebellar ataxia. The ICARS is a 0- 100 point scale system with four subscales that include, postural and gait disturbances, limb ataxia, dysarthria, and Oculomotor disorders. Postural and gait disturbances are scaled 0 to 34 points. Limb ataxia is scaled 0 to 52 points. Dysarthria is scaled 0 to 8 points, and Oculomotor disorders is scaled 0 to 6 points. The higher the score indicates greater impairment.
ARAT ( Action Research Arm Test) | Assessed week 1 before the first training session, and week 12
  The ARAT is an assessment used to measure changes in upper limb function in people who have experienced damage or disease to the nervous system (e.g., multiple sclerosis, stroke, Parkinson's disease, cerebellar ataxia).

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Bastian, PhD, PT, Principal Investigator — Kennedy Krieger Institute and Johns Hopkins School of Medicine
Locations (1):
- Motion Analysis Lab in the Kennedy Krieger Institute, Baltimore, Maryland, United States